CLINICAL TRIAL: NCT04611373
Title: A Single-center, Single-arm, Open, Prospective, and Exploratory Clinical Study on the Efficacy of Acetazolamide Combined With Levamisole in the Treatment of Advanced HCC
Brief Title: Clinical Study on the Efficacy of Acetazolamide Combined With Levamisole in the Treatment of HCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Zujiang YU, The First Affiliated Hospital of Zhengzhou University, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CJVICC-001
Record Dates: First submitted 2020-10-28; First posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: HCC

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A (Experimental): Acetazolamide tablet 25mg/ tablet, 2 tablets a day; Levamisole 25mg/ tablet, 6 tablets/day continuous medication; Continue treatment until the disease progresses
  Interventions: Drug: Acetazolamide Levamisole

INTERVENTIONS:
Drug: Acetazolamide Levamisole — Acetazolamide tablet 25mg/ tablet, 2 tablets a day Levamisole 25mg/ tablet, 6 tablets/day Continue treatment until the disease progresses

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of acetazolamide combined with levamisole in the treatment of advanced HCC.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the sixth most common cancer and the second leading cause of cancer-related deaths in the world. Because HCC is insidious and early diagnosis is difficult, most patients have locally advanced or distant metastasis at the time of diagnosis. So they are not suitable candidates for curative treatments by resection or transplantation. Currently, There are only not more than five drugs to be selected for advanced HCC, although it prolongs the survival for less than 3 months. Recently, metabolomics studies of HCC have shown that typical Warburg effect was observed in hepatoma carcinoma cells. Arginine hydrochloride is a new anticancer drug in the treatment of HCC, which is mainly aimed at the pathway of energy metabolism.acetazolamide may play an anti-tumor role by inhibiting the reverse TCA cycle. The investigators have been proceeding this trial to evaluate the efficacy and safety of acetazolamide combined with levamisole in the treatment of advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-65 years
2. The diagnosis of ICC: in accordance with "diagnostic and treating standards on primary liver cancer" or histological/cytological diagnosis of primary liver cancer
3. Un-resectable HCC : patients with developing primary liver cancer of Barcelona stage(BCLC) B; multiple nodules (less than 5, the total diameter of less than 20 cm), no invasion, no symptoms;refusing open surgical treatment and volunteering for the treatment
4. The First-line system therapy failure (or residual lesion) from the group of this study a signed informed consent (time) for 2 weeks or more basic returned to normal and adverse events (NCI CTCAE Ⅰ level or less);
5. Child-Pugh liver function class A/B(score: ≤7)
6. Performance status 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale in one week before admission
7. Estimated survival time > 3 months
8. HBV DNA#2000 IU/ml#10^4 copies/ml); or HBV DNA≥2000 IU/ml and are accepting effective antiviral therapy
9. The major organ function is normal. that is meeting the following standards:

   Blood routine examination: (No blood transfusion, no G-CSF and no medication were corrected within 14 days before screening)
10. For women of childbearing age, the results of serum/urine pregnancy tests must be negative within 7 days before initiation of treatment. All men and women who participate in the study have to take reliable contraceptive measures within the trial and eight weeks after the trial is completed
11. volunteers must signed informed consent

Exclusion Criteria:

1. With a history of alimentary tract hemorrhage or a definite tendency of gastrointestinal bleeding, such as varices of fundus of stomach and esophagus with bleeding risk; local active ulcer lesions; fecal occult blood ≥#++#
2. Patients with hepatobiliary cell carcinoma, mixed cell carcinoma or lamellar cell carcinoma; in the past (within 5 years) or at the same time suffering from other untreated malignant tumors; excluding cured basal cell carcinoma and carcinoma in situs of cervix
3. Patients who are undergoing liver transplantation or have a history of organ transplantation(excluding the patient who has undergone liver transplantation before)
4. Patients with an allergic history of Levamisole Hydrochloride and Anlotinib Hydrochloride Capsules
5. The blood pressure can not be reduced to the normal range by the antihypertensive drug treatment in patients with hypertension(systolic pressure#140 mmHg, diastolic pressure#90 mmHg)
6. Patients with myocardial ischemia or myocardial infarction over grade II or a poorly controlled arrhythmia (including QTc interval: men ≥ 450 ms; women ≥ 470 ms)
7. Cardiac functional insufficiency of grade III to IV according to NYHA standard; echocardiography: LVEF#50%
8. Many factors that influence oral medication, such as unable to swallow; chronic diarrhea; intestinal obstruction; the situations which significantly affect the use and absorption of drugs
9. Abdominal fistula, gastrointestinal perforation, or abdominal abscess occurred within 28 days before participating the study
10. Dysfunction of blood coagulation(INR#2.0 or PT# 16s#APTT > 43s#TT > 21s#Fbg < 2g/L), having a tendency to bleed or undergoing thrombolysis or anticoagulant therapy; ascites with clinical symptoms, that is requiring therapeutic abdominal paracentesis or drainage or Child-Pugh score ≥2
11. Objective evidence of pulmonary fibrosis history, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug associated pneumonia, and severe lung function impairment in the past and at present
12. Urine routine showed that urine protein ≥++ or the urine protein in 24 hours#1.0 g
13. Patients who have been treated with potent CYP3A4 inhibitors (ketoconazole, itraconazole, voriconazole, ritonavir, clarithromycin, telithromycin, troleandomycin, erythromycin, cimetidine and so on) within 28 days before participating the study, or potent CYP3A4 inducers (dexamethasone, phenytoin, rifampin, rifabutin, carbamazepine, phenobarbitone and so on) within 12 days before participating the study.
14. Pregnant or lactating women; fertile patients who are unwilling or unable to adopt effective contraceptives
15. Patients with mental sickness or the history of psychotropic drug abuse
16. Patients with severe infection (unable to control the infection effectively)
17. The treatment history affecting this program or its efficacy, such as stem cell transplantation, immune regulation (including PD-1 and other test regimens) recently (within half a year)
18. The researchers believe that any other factors unsuitable for entering into the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | 24 months
  Time from start of treatment until the first documented event of symptomatic progression or death

SECONDARY OUTCOMES:
Overall Surviva | 48 months
  ime from start of treatment to death from any cause, or last known date of survival

OTHER OUTCOMES:
Disease Control Rate(DCR) | 28 days
  the percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease
Objective Response Rate(ORR) | 28 days
  Proportion of patients with reduction in tumor burden of a predefined amount
The change of AFP biomarker | 28 days
  Concentration of AFP biomarker change in tumor markers

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No